CLINICAL TRIAL: NCT01257750
Title: Safety and Efficacy of Topical Pazopanib in Treatment of Corneal Neovascularization
Brief Title: Treatment of Corneal Neovascularization With Topical Pazopanib
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Reza Dana, MD (Other)
Responsible Party: Sponsor-Investigator, Reza Dana, MD, Principal Investigator, Massachusetts Eye and Ear Infirmary
Organization: Massachusetts Eye and Ear Infirmary (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-09-063
Record Dates: First submitted 2010-11-22; First posted 2010-12-10 (Estimated); Results first posted 2012-11-06 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2017-12

CONDITIONS: Corneal Neovascularization
Keywords: corneal neovascularization; pazopanib; votrient; rosacea
MeSH Terms: conditions — Corneal Neovascularization; Rosacea | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pazopanib (Experimental): This is a single site, open label, safety and efficacy study of pazopanib (5mg/ml) where all 20 patients with corneal neovascularization in a single arm will receive pazopanib in one eye.
  Interventions: Drug: Pazopanib (5mg/ml)

INTERVENTIONS:
Drug: Pazopanib (5mg/ml) — Topical pazopanib, 4 times per day for 3 weeks
  Other Names: Votrient

SUMMARY:
The purpose of this study is to determine the safety and efficacy of a drug [Pazopanib (Votrient)] as a treatment for corneal neovascularization. The cornea is the clear, central portion of the eye and neovascularization means blood vessel growth. The cornea is typically avascular, or without blood vessels. Corneal neovascularization in the cornea and can put vision at risk. Numerous diseases of the cornea such as inflammation, ischemia (restriction of blood supply), infection, degeneration (or deterioration), trauma, or corneal stem cell deficiency can lead to corneal neovascularization. This major ocular complication can lead to corneal scarring, edema (swelling), lipid deposits, and inflammation that may significantly alter your vision. In addition, it worsens the outcome of potential future treatments, such as a corneal transplant. A corneal transplant is a treatment that many patients with severe corneal disease may ultimately need.

DETAILED DESCRIPTION:
Normally avascular, under many pathologic conditions, vessels may invade the cornea from the limbal vascular plexus. Infection, inflammation, ischemia, degeneration, or trauma, and the loss of the limbal stem cell barrier can cause corneal neovascularization. Growth of new vessels may result in corneal scarring, edema, lipid deposition, and inflammation that may alter visual acuity and is a leading cause of monocular visual impairment and blindness. Additionally, it results in the loss of immune response across the cornea, thereby worsening the prognosis of a subsequent penetrating keratoplasty (PK). Growth of new blood and lymphatic vessels from preexisting vessels are mediated by members of the vascular endothelial growth factor (VEGF) family. In previous studies, inhibition of new blood or lymphatic vessels has been achieved by neutralization of vascular endothelial growth factor A (VEGF-A). It has also been shown that platelet-derived growth factor-B (PDGF-B) plays a role in corneal and choroidal neovascularization by regulating mural cell recruitment. Inhibition of PDGF-B and VEGF-A signaling pathways has shown to more effectively promote vessel regression than solely inhibiting VEGF-A. Pazopanib is a drug designed to block these pathways, stop new growth, and regress old vessel growth.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Ability to comply with study assessments and study requirements (for example, able to open the eye drop foil-wrap packaging and eye drop vials, willing to adhere to the daily dosing schedule) for the full duration of study
* Age > 18 years
* Patients with superficial or deep corneal neovascularization that extends farther than 1 mm from the limbus
* Patients are in stable overall health
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase and bilirubin ≤ 1.5x upper limit of normal (ULN) or isolated bilirubin >1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%
* Single QTcF < 450 msec; or QTcF < 480 msec in subjects with Bundle Branch Block
* A female is eligible to enter and participate in this study if she is of Non-childbearing potential (i.e., physiologically incapable of becoming pregnant),

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* History of any clotting disorder, including predisposition to hypercoagulation or any previous thromboembolic event
* Major surgery within 1 month of screening
* Has received treatment with anti-VEGF agents (topical, intraocular or systemic) within 60 days of study entry. This includes both approved and investigational treatments.
* Has received investigational therapy within 60 days prior to study entry
* Concurrent enrollment in another clinical investigational medicinal product or device study
* Concurrent use of anti-VEGF agents
* Corneal or ocular surface infection within 30 days prior to study entry
* Full thickness or lamellar keratoplasty within 90 days prior to study entry
* Other ocular surgeries within 60 days prior to study entry
* Ocular or periocular malignancy
* Soft Contact lens (excluding bandage contact lens) use within 2 weeks prior to study entry
* Persistent epithelial defect (>1mm and ≥14 days duration) within 2 weeks prior to study entry
* Intravitreal or periocular steroids within 4 weeks prior to study entry
* Change in dose/frequency of topical steroids and/or nonsteroidal anti-inflammatory drugs (NSAIDs) within 2 weeks prior to study entry
* Poorly controlled Hypertension: systolic blood pressure (BP) > 150 or diastolic BP > 90
* Medical history of uncontrolled diabetes mellitus, with hemoglobin A1c (HbA1c) >7%
* Women 45 years of age or younger that are of child bearing potential as defined by:

  * No history of a hysterectomy
  * No history of a bilateral oophorectomy (ovariectomy)
  * No history of a bilateral tubal ligation
  * Not post-menopausal
* Subjects using hormone replacement therapy (HRT) that have experienced total cessation of menses for ≤ 1 year, OR, in questionable cases, have a follicle stimulating hormone (FSH) value <40 mIU/mL and an estradiol value > 40pg/mL (>140 pmol/L) OR have documented evidence OR have had documented evidence of menopause based on FSH and estradiol concentrations prior to initiation of HRT. Signs of current infection, including fever and current treatment with antibiotics
* Participation in another simultaneous medical investigation or trial STUDY

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reza Dana, MD, MPH, MSc, Principal Investigator — Mass Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Amparo F, Sadrai Z, Jin Y, Alfonso-Bartolozzi B, Wang H, Shikari H, Ciolino JB, Chodosh J, Jurkunas U, Schaumberg DA, Dana R. Safety and efficacy of the multitargeted receptor kinase inhibitor pazopanib in the treatment of corneal neovascularization. Invest Ophthalmol Vis Sci. 2013 Jan 17;54(1):537-44. doi: 10.1167/iovs.12-11032. PMID 23233252

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited and consented at the Massachusetts Eye and Ear Infirmary Cornea Department from November 2010 - October 2011.
Groups:
- Pazopanib: This is a single site, open label, safety and efficacy study of pazopanib (5mg/ml) where all 20 patients with corneal neovascularization in a single arm will receive pazopanib in one eye.
  Frequency and Duration: 4 times per day for 3 weeks
Period: Overall Study
Arm/Group | Pazopanib
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pazopanib
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 20
Mean Arterial Pressure [Mean (Standard Deviation); unit: mm Hg] | 92.0 (1.7)
Heart Rate [Mean (Standard Deviation); unit: Beats per Minute] | 70.4 (8.1)
Intraocular Pressure [Mean (Standard Deviation); unit: mm Hg] | 15.7 (5.9)
Central Corneal Thickness [Mean (Standard Deviation); unit: microns] — Corneal pachymetry is used to measure central corneal thickness. This technique is used to gauge the functional status of the corneal endothelial cell layer.
  microns | 572 (135)

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate
Description: Heart rate through was measured throughout the study to assess subjects for systemic adverse events.
Time Frame: 12 Weeks
Population: All enrolled patients were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per Minutes
Arm/Group | Pazopanib
Number analyzed (Participants) | 20
Beats per Minutes | 68.7 (7.6)

2. Primary Outcome: Mean Arterial Pressure
Description: Mean arterial pressure was measured throughout the study to assess subjects for systemic adverse events..
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Pazopanib
Number analyzed (Participants) | 20
mmHG | 90.7 (1.4)

3. Primary Outcome: Central Corneal Thickness
Description: Pachymetry was used to measure the central corneal thickness of each study subject. Central corneal thickness was measured throughout the study to assess subjects for ocular adverse events.
Time Frame: 12 Weeks
Population: All enrolled patients were analyzed.
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Pazopanib
Number analyzed (Participants) | 20
Microns | 590 (162)

4. Primary Outcome: Intaocular Pressure
Description: Intaocular pressure is the measurement of pressure within the eye. Intaocular pressure was measured throughout the study to assess subjects for ocular adverse events.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Pazopanib
Number analyzed (Participants) | 20
mmHg | 16.9 (5.3)

5. Secondary Outcome: Corneal Neovascular Area
Description: Corneal neovascular area is the measurement of the area of the cornea where new blood vessels are forming. The mean Change in Corneal Neovascular Area from Baseline to 12 Week Time Point is reported below.
Time Frame: Through 12 weeks of Follow-Up
Population: Mean Change in Corneal Neovascular Area (measuring the area of the corneal vessels) from Baseline to 12 Week Time Point.
Measure: Mean (Standard Deviation); unit: millimeters squared
Arm/Group | Pazopanib
Number analyzed (Participants) | 20
millimeters squared | 1.5 (0.8)

6. Secondary Outcome: Corneal Invasion Area
Description: Corneal Invasion area is the measurement of the fraction of the total corneal area that is invaded by blood vessels. The mean Change in Corneal invasion area from baseline to 12 Week Time Point is reported below.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: millimeters squared
Arm/Group | Pazopanib
Number analyzed (Participants) | 20
millimeters squared | 3.9 (1.8)

7. Secondary Outcome: Corneal Vessel Length
Description: Corneal vessel length is the measurement of the length of the extent of vessels from end to end. The mean change in corneal vessel length from Baseline to 12 Week Time Point is reported below.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Pazopanib
Number analyzed (Participants) | 20
millimeters | 38.0 (17.2)

8. Secondary Outcome: Corneal Vessel Caliber
Description: Corneal vessel caliber is the measurement of the diameter of the corneal blood vessels. The mean change in the corneal vessel caliber from baseline to 12 week time point is reported below.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Pazopanib
Number analyzed (Participants) | 20
millimeters | 0.0003 (0.0005)

ADVERSE EVENTS:
Arm/Group | Pazopanib
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 12/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pazopanib (N=20)
Tearing (Eye disorders) | 10 (13) — Unilateral tearing secondary to punctal occlusion.
Stinging (Eye disorders) | 4 (4) — Transitory stinging directly related to drug instillation.
Dryness (Eye disorders) | 1 (1)
Blurred Vision (Eye disorders) | 1 (1) — Blurred vision after drug instillation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes